CLINICAL TRIAL: NCT04493788
Title: Novel Molecular Characterization of Oocytes and Cumulus Cells From Women With Polycystic Ovarian Syndrome (PCOS) Phenotype A
Brief Title: Molecular Basis of PCOS in Oocytes and Surrounding Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: MOLPA-2020253
Record Dates: First submitted 2020-07-20; First posted 2020-07-30 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Hematologic Tests; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS group
  Interventions: Other: Blood test, ultrasound and egg retrieval
- Control group
  Interventions: Other: Blood test, ultrasound and egg retrieval

INTERVENTIONS:
Other: Blood test, ultrasound and egg retrieval — Blood tests will be performed to determine free testosterone levels, anti-mullerian hormone (AMH) and lipid profile including fasting plasma glucose and insulin. Women from both PCOS and control groups will be minimally stimulated with gonadotrophins and cumulus-oocytes complexes (COCs) will be aspirated from small antral follicles (2-8mm) without any ovulation triggering. Specifically, administration of highly purified human menopausal gonadotropin (HP-hMG) will start on cycle Day 3 of the menstrual period or a withdrawal bleeding. A pelvic ultrasound scan will be performed in the morning of the last stimulation day to schedule the oocyte collection. Cumulus-oocyte complexes retrieved 42 hours after the last gonadotropin injection will be collected, washed, denuded and individually stored for further molecular characterization.

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common disorder in women of reproductive age that is characterized by elevated androgen levels, ovulatory dysfunction and polycystic ovarian morphology (PCOM). Moreover, has been associated to insulin resistance, obesity, type 2 diabetes and infertility.

Women with PCOS are a heterogeneous group, and specific PCOS phenotype could have a substantial impact on oocyte quality and molecular profile. Regarding the Rotterdam criteria for PCOS, four different phenotypes of the syndrome are defined (A, B, C, D). Phenotypic group A is the most frequent and severe subtype of PCOS. It is described that patients with so-called phenotype A exhibit a significantly increased risk of pregnancy complications compared to women with more favorable PCOS phenotypes. Specifically, this clinical-laboratory study will focus on the molecular characterization of PCOS phenotype A.

Epigenetic are external modifications to DNA that affect how cells "read" genes. These external modifications have garnered attention in the pathogenesis of PCOS since epigenetics changes have been reported in various organs in women with the condition. However, remains unknown whether these alterations are also found in the egg and in its surrounding cells.

Further research is needed to understand the PCOS disorder and to design treatments that can ameliorate the symptoms of the disease. In particular, this project aims to generate the molecular profiles of PCOS phenotype A eggs and surrounding cells and compare them with the ones obtained from and healthy controls. This approach involves the aspiration of immature eggs without hormonal stimulation or with stimulation of only a few days.

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 18 and 37
* biochemical hyperandrogenism
* ovulatory dysfunction
* polycystic ovaries)
* BMI > 25.
* normal andro-gen levels
* normal ovarian function
* normal ovarian morphology
* BMI < 29.

Exclusion Criteria:

* congenital adrenal hyperplasia
* Cushing's syndrome
* androgenic-secreting tumor
* high (>grade 2) grade endometriosis
* major uterine or ovarian abnormalities
* pregnant women
* volunteers with metabolic syndrome

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Research material will be collected from (i) PCOS patients with phenotype A undergoing IVM who donate part of their oocytes for research, and (ii) women with normal ovaries and androgen levels who also donate the total amount of the retrieved oocytes for research. Participants between the ages of 18 and 37 will be enrolled through correspondent recruitment programs running in the Centre for Reproductive Medicine of UZ Brussel (CRG). BMI will be determined and blood tests will be performed to determine free testosterone levels, AMH and lipid profile including fasting plasma glucose and insulin. The PCOS group will include patients with phenotype A and the age-matched control groups will include volunteers with normal androgen levels.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
DNA methylation profiles in oocytes and cumulus cells | This information is expected to be generated in 24 months
  On of the primary outcome measure of this project will be the generation of DNA methylation profile of PCOS oocytes and paired cumulus cells using single-cell and low-cell parallel sequencing, respectively.
Gene expression profiles in oocytes and cumulus cells | This information is expected to be generated in 24 months
  Another primary outcome measure of this project will be the generation of gene expression profile of PCOS oocytes and paired cumulus cells using single-cell and low-cell parallel sequencing, respectively.